CLINICAL TRIAL: NCT01638572
Title: Exploring the Possibility to Use Glycosyltransferase as a Prognosis Marker of Neuroblastoma
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200910002R
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; B4GALNT3; Prognosis
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- neuroblastoma patients

SUMMARY:
Well-regulated glycosylation is essential for the normal development of the nervous system. Altered expression of glycosyltransferases with resulting dysregulated glycosylation of neuroblastic cells might lead to the development of NB. The β1,4-N-acetylgalactosaminyltransferase III (B4GALNT3) exhibits GalNAc transferase activity to form the GalNAcβ1,4GlcNAc (LacdiNAc or LDN) structure. The Drosophila B4GALNTA, homolog of human B4GALNT3, has been suggested to regulate the neuronal development. By immunohistochemical studies, we demonstrated that the expression of B4GALNT3 correlated well with histological grade of differentiation in NB tumor samples. Since well differentiated tumors usually carry a better prognosis, we thus speculate that expression of B4GALNT3 in tumor tissues can a favorable prognostic factor of NB.

To explore the role of B4GALNT3 in the prognosis of NB, we propose the following project with two specific aims:

Aim Ⅰ: Establishing the significance of B4GALNT3 in the prognosis of NB: We plan to collect 90 NB tumor samples, and evaluate the RNA and protein expression levels by Q-PCR, Western blot, and immunohistochemistry in the tumor samples. The results will be compared with the other clinicopathological and biological factors of NB. Also the expression levels of B4GALNT3 in tumor tissues will be correlated to the patients' outcome to clarify whether B4GALNT3 could be a prognosis marker of NB.

Aim II: Clarifying the effects of B4GALNT3 on NB cell behavior in vitro and in vivo. For further strengthening the prognostic role of B4GALNT3 in NB, NB cell phenotype and behavior changes after overexpression or knock-down of B4GALNT3 are evaluated by in vitro assays as well as by a nude mice xenograft model.

In summary, if our project can establish the role of B4GALNT3 expression in NB, we may further subclassify the NB patients, and give the NB patients more appropriate therapies to improve patients' outcome. Furthermore, B4GALNT3 could potentially serves as a therapeutic target in the future.

ELIGIBILITY:
Inclusion Criteria:

* Neuroblastoma patients with complete follow-up and sufficient samples for study

Exclusion Criteria:

* Neuroblastoma patients without complete follow-up or sufficient samples for study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: From year 1990 to 2010, pediatric neuroblastoma patients treated at National University Hospital, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ming Hsu, M.D, Ph.D, Principal Investigator — National Taiwan Univesity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan